CLINICAL TRIAL: NCT07162519
Title: A Prospective, Single-arm, Multicenter Clinical Study of Romiplostim N01 in the Treatment of Thrombocytopenia Caused by Cytotoxic Drugs in Breast Cancer Patients.
Brief Title: Romiplostim N01 in the Treatment of Thrombocytopenia Caused by Cytotoxic Drugs in Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Affiliated Hospital of Hebei University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shandong Cancer Hospital and Institute (Other); Tangshan People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-CTIT-RULS-1002
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Cytotoxic Drugs; Romiplostim N01; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug Intervention Group - Treated with Romiplostim N01 (Experimental)
  Interventions: Drug: romiplostim N01

INTERVENTIONS:
Drug: romiplostim N01 — Eligible subjects who pass the screening will undergo a baseline visit and will receive romiplostim N01 administration once weekly for a maximum of 4 weeks. Dosing will be discontinued when the platelet count rises to ≥100×10⁹/L. When a subject resumes anti-tumor therapy, those with a baseline platelet count of <50×10⁹/L will receive prophylactic administration of romiplostim N01 (administered 2 hours prior to anti-tumor therapy) before the anti-tumor drugs are given.

SUMMARY:
The primary study objective:

To evaluate the efficacy of romiplostim (N01) in the treatment of chemotherapy-induced thrombocytopenia (CIT) in breast cancer patients by assessing the proportion of patients whose platelet count recovers to ≥100×10⁹/L after two weeks of treatment.

This study is a multicenter, single-arm, interventional trial. It plans to enroll 68 breast cancer patients with chemotherapy-induced thrombocytopenia (CIT) (PLT <75×10⁹/L).

The study comprises a Screening Period (from after the subject signs the informed consent form until before the first dose), a Treatment Period (including treatment with romiplostim N01), and a Follow-up Period.

Screening Period: Subjects will be evaluated against the inclusion and exclusion criteria. Those who qualify may proceed to the Treatment Period.

Treatment Period: Eligible subjects from screening will undergo a baseline visit and will receive romiplostim N01 once weekly for a maximum of 4 weeks. Dosing will be stopped when the platelet count increases to ≥100×10⁹/L. When a subject resumes anti-tumor therapy, prophylactic administration of romiplostim N01 (administered 2 hours prior to anti-tumor therapy) will be performed for subjects with a baseline platelet level of <50×10⁹/L before the administration of the anti-tumor therapy drugs.

Dosage Regimen:

Romiplostim N01: 200 μg per dose, administered subcutaneously, once weekly.

Follow-up Period: Subjects will enter the Follow-up Period after the completion of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained prior to enrollment;
2. Aged 18-75 years;
3. Patients with histologically or pathologically confirmed breast cancer;
4. Breast cancer patients with chemotherapy-induced thrombocytopenia (CTIT);
5. No prior treatment with romiplostim or romiplostim N01 within 3 months;
6. ECOG PS score: 0-2;
7. Platelet count <75×10⁹/L;
8. Expected survival period ≥12 weeks at screening;
9. Subjects of childbearing potential must agree to use reliable contraception throughout the study period (including male or female condoms, contraceptive foam, gel, film, cream, suppositories, abstinence, or intrauterine devices, etc.). Exceptions include female subjects who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation, or postmenopausal status for over 1 year, and male subjects who have undergone bilateral vasectomy or ligation;
10. Voluntarily participate in the study, sign informed consent, and demonstrate good compliance.

Exclusion Criteria:

1. Presence of hematopoietic system diseases other than chemotherapy-induced thrombocytopenia (CIT), including but not limited to leukemia, primary immune thrombocytopenia, myeloproliferative disorders, multiple myeloma, and myelodysplastic syndromes;
2. Platelet reduction due to causes other than CIT within 6 months prior to screening, including but not limited to chronic liver disease, hypersplenism, infection, or hemorrhage;
3. Bone marrow infiltration or bone marrow metastasis;
4. Prior radiotherapy to the pelvis, spine, or large-field bone irradiation within 3 months before screening, or current/scheduled radiotherapy;
5. History of severe cardiovascular diseases within 6 months prior to screening, such as congestive heart failure (NYHA Class III-IV), arrhythmias known to increase thromboembolic risk (e.g., atrial fibrillation), post-coronary stent implantation, angioplasty, or coronary artery bypass grafting;
6. Clinical manifestations of severe hemorrhage within 2 weeks before screening, such as gastrointestinal or central nervous system bleeding;
7. Brain tumors or brain metastases;
8. Conditions requiring emergency treatment, such as superior vena cava syndrome or spinal cord compression;
9. Absolute neutrophil count <1.0×10⁹/L or hemoglobin <80 g/L (use of granulocyte colony-stimulating factor, red blood cell transfusions, or EPO therapy per clinical practice is allowed);
10. Significant liver dysfunction: For patients without liver metastases, ALT/AST >3×ULN (upper limit of normal) or TBIL >3×ULN; for patients with liver metastases, ALT/AST ≥5×ULN or TBIL ≥5×ULN;
11. Renal dysfunction: Serum creatinine ≥1.5×ULN or eGFR ≤60 mL/min (calculated by Cockcroft-Gault formula);
12. Known or expected hypersensitivity or intolerance to romiplostim N01 or excipients of rhTPO; 13．HIV-infected patients; 14．Pregnant or lactating women; 15．Participation in any other clinical trial involving investigational drugs or devices within 3 months prior to screening; 16．Other situations deemed by the investigator to pose significant risks to the subject's health or safety, or potentially affecting efficacy evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
2-week response rate | 2 weeks
  The proportion of patients whose platelet count recovers to ≥100×10⁹/L within 2 weeks of treatment.

SECONDARY OUTCOMES:
The median time for platelet count to recover to ≥75×10⁹/L after treatment; | 1 month
  The median time for platelet count to recover to ≥75×10⁹/L after treatment;
The proportion of patients achieving a platelet count recovery to ≥75×10⁹/L within 2 weeks of treatment. | 2 weeks
  The proportion of patients achieving a platelet count recovery to ≥75×10⁹/L within 2 weeks of treatment.
The absolute value of the change in platelet count from baseline within 2 weeks of treatment. | 1 month
  The absolute value of the change in platelet count from baseline within 2 weeks of treatment.
The proportion of patients achieving an increase in platelet count of ≥30×10⁹/L from baseline within 2 weeks of treatment. | 2 weeks
  The proportion of patients achieving an increase in platelet count of ≥30×10⁹/L from baseline within 2 weeks of treatment.
The median time to platelet count recovery to ≥100×10⁹/L following treatment initiation. | 1 month
  The median time to platelet count recovery to ≥100×10⁹/L following treatment initiation.
The proportion of patients who resumed antitumor therapy within two weeks. | 2 weeks
  The proportion of patients who resumed antitumor therapy within two weeks.
The maximum platelet count within two weeks of treatment. | 2 weeks
  The maximum platelet count within two weeks of treatment.
The number of platelet transfusions and the transfusion volume during the study period. | 1 month
  The number of platelet transfusions and the transfusion volume during the study period.
The proportion of patients with a dose reduction of cytotoxic drugs by ≥15% due to CTIT following secondary prophylaxis. | 1 month
  The proportion of patients with a dose reduction of cytotoxic drugs by ≥15% due to CTIT following secondary prophylaxis.
The proportion of patients who developed CTIT after secondary prophylaxis. | 1 month
  The proportion of patients who developed CTIT after secondary prophylaxis.

IPD SHARING:
Plan to Share IPD: Undecided